CLINICAL TRIAL: NCT00650637
Title: A Randomized, Open-Label, Third-Party Blinded Study for the Prophylaxis and Treatment of Nelfinavir-associated Diarrhea
Brief Title: A Study to Determine Effective Prophylaxis and Treatment of Nelfinavir-Associated Diarrhea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to administrative reasons on August 18, 2003. There were no safety concerns that led to the decision to terminate.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A4301004
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Calcium Carbonate; Nelfinavir; Lamivudine; Loperamide; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Calcium Carbonate; Drug: nelfinavir; Drug: lamivudine; Drug: loperamide
- 2 (Experimental)
  Interventions: Other: Calcium carbonate not administered; Drug: nelfinavir; Drug: lamivudine + zidovudine

INTERVENTIONS:
Drug: Calcium Carbonate — Calcium carbonate 500 mg oral tablet twice a day; given in combination with the following antiretroviral combination: nelfinavir 1250 mg twice a day, and lamivudine 150 mg/zidovudine 300 mg twice a day (or stavudine 40 mg twice a day plus lamivudine 150 mg twice a day); If diarrhea develops, loperamide 2 mg oral caplet 3 times weekly; All study drugs continued through to Week 12
  Arms: 1
Drug: nelfinavir — 1250 mg twice a day
  Other Names: Viracept
  Arms: 1
Drug: lamivudine — lamivudine 150 mg/zidovudine 300 mg twice a day (or stavudine 40 mg twice a day plus lamivudine 150 mg twice a day);
  Arms: 1
Drug: loperamide — If diarrhea develops, loperamide 2 mg oral caplet 3 times weekly;
  Arms: 1
Other: Calcium carbonate not administered — Prophylaxis with calcium carbonate not administered in this group; The following antiretroviral combination was administered: nelfinavir 1250 mg twice a day, and lamivudine 150 mg/zidovudine 300 mg twice a day (or stavudine 40 mg twice a day plus lamivudine 150 mg twice a day);
  Arms: 2
Drug: nelfinavir — nelfinavir 1250 mg twice a day
  Other Names: Viracept
  Arms: 2
Drug: lamivudine + zidovudine — lamivudine 150 mg/zidovudine 300 mg twice a day (or stavudine 40 mg twice a day plus lamivudine 150 mg twice a day);
  Arms: 2

SUMMARY:
The purpose of this study was to determine the efficacy and safety of calcium carbonate for the prevention of nelfinavir-associated diarrhea and to evaluate the efficacy and safety of calcium carbonate in combination with loperamide for the treatment of nelfinavir-associated diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral-naive patients with HIV-1 infection
* not more than 2 loose stools per day or any preexisting or emerging medical condition that would interfere with the evaluation of therapeutic response of the study drug
* No antidiarrheal medication within 7 days prior to entry

Exclusion Criteria:

* Greater than or equal to 2 loose stools per day lasting 2 or more days within 7 days prior to study entry
* Bloody stools within 7 days prior to study entry
* Any unstable or severe intercurrent medical condition, including active opportunistic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-01; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Number of patients who experienced protocol-defined diarrhea in each treatment group during study | Week 12

SECONDARY OUTCOMES:
Time to first occurrence of protocol-defined diarrhea
The outcome of calcium carbonate plus loperamide in treating subjects who experienced diarrhea | Weeks 2, 4, 6, 8, and 12
Frequency and severity of diarrhea collected from the subject daily diary during the study will be summarized before and after subjects receive calcium carbonate plus loperamide | Weeks 2, 4, 6, 8, and 12
Safety evaluations including physical exam, weight and vital signs measurements | Screening, baseline, Weeks 2, 4, 6, 8, and 12
Safety assessment of laboratory parameters | Screening, baseline, Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4301004&StudyName=A%20Study%20to%20Determine%20Effective%20Prophylaxis%20and%20Treatment%20of%20Nelfinavir-Associated%20Diarrhea.